CLINICAL TRIAL: NCT02732496
Title: Computerized Working Memory Training in Children With Attention-Deficit/Hyperactivity Disorder and Comorbid Tourette Syndrome
Brief Title: Computerized Working Memory Training in Children With ADHD and Comorbid Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Louis V. Gerstner III Research Scholar Award (Unknown)
Responsible Party: Principal Investigator, Mary Zelime Elibol, Instructor in Neurology, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P002512
Record Dates: First submitted 2016-03-03; First posted 2016-04-08 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; Tourette Syndrome
Keywords: Attention-Deficit/Hyperactivity Disorder; Tourette Syndrome; Working Memory Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Experimental): Targeted Cognitive Training (TCT)
  Interventions: Behavioral: Targeted Cognitive Training (TCT)
- Youth Appropriate Online Games (Placebo Comparator): Engaging games not designed to improve cognition
  Interventions: Other: Youth Appropriate Online Games

INTERVENTIONS:
Behavioral: Targeted Cognitive Training (TCT) — The instructors have selected a set of computer exercises designed to specifically target working memory, which is a cognitive construct relevant to ADHD and Tourette Syndrome. The tasks were designed to benefit subjects through principles of learning-dependent plasticity.
  Arms: Cognitive Training
Other: Youth Appropriate Online Games — Engaging games not designed to improve cognition.
  Arms: Youth Appropriate Online Games

SUMMARY:
The investigators will conduct a randomized placebo-controlled trial of a computerized intervention targeting working memory in 30 children with comorbid Attention-Deficit/Hyperactivity Disorder (ADHD) and Tourette Syndrome (TS).

DETAILED DESCRIPTION:
Because impairments in executive functions (EFs), such as working memory, are associated with functional impairments in youth with neurodevelopmental and neuropsychiatric disorders, strategies that target EFs are critical. Neuroplasticity-based cognitive training has been found to improve cognition in youth with ADHD and in adults with schizophrenia. In this trial, the investigators seek to extend the relevance of computerized cognitive training to youth with comorbid ADHD and Tourette Syndrome. Given the literature, the investigators hypothesize that computerized working memory training will produce gains in untrained cognitive tasks and behavioral ratings of executive functions in youth with ADHD+TS. The investigators will assess aspects of attention and executive functions in 30 affected youth and randomize them 1:1 to either neuroplasticity-based cognitive training or enjoyable age-appropriate computer games not intended to improve cognition. Cognition will be assessed again after 30 training sessions over 6 weeks and then again at a one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The investigators will limit inclusion to youth between the ages of 7-13 who carry current diagnoses of ADHD+TS and who have a treating physician at a Partners affiliated hospital or clinic.
2. The investigators will include youth who have undergone neuropsychological testing in the prior 3 years.

Exclusion Criteria:

1. The investigators will exclude patients with intellectual disability in order to more directly extend the prior literature to the ADHD+TS population.
2. The investigators will exclude patients with severe tics as evidenced by a score of > 30 on the clinician administered Yale Global Tic Severity Scale (YGTSS).
3. The investigators will exclude patients with moderate to severe Obsessive Compulsive Disorder (OCD) symptoms, as evidenced by a score of >30 on the clinician administered Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS).
4. The investigators will exclude patients treated with neuroleptics, given that these medications can be cognitively dulling and sedating and potentially lead to secondary working memory impairments.
5. The investigators will exclude families who do not have a computer with an internet connection in their homes, and in which neither a parent nor the child has an email address to receive study related communications.
6. The investigators will exclude families who anticipate or are likely to have a change in therapeutic treatments (i.e., psychotherapy or psychopharmacology) during the time frame of the trial.

NOTE: Patients treated with ADHD medications will not be excluded, but medications will be recorded for covariate analysis.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Spatial Working Memory (SWM) subtest from the Cambridge Neuropsychological Test Automated Battery (CANTAB) | 3 months
  The SWM subtest assesses working memory.
Spatial Span (SSP) subtest from the Cambridge Neuropsychological Test Automated Battery (CANTAB) | 3 months
  The SSP subtest assesses working memory.
The Working Memory Index from the Behavior Rating Inventory of Executive Function (BRIEF) | 3 months
  Parent and teacher ratings on the Working Memory Index of the BRIEF assess working memory.
The Behavioral Regulation Index from the Behavior Rating Inventory of Executive Function (BRIEF) | 3 months
  Parent and teacher ratings on the Behavioral Regulation Index of the BRIEF assess working memory.

CONTACTS AND LOCATIONS:
Overall Officials: M. Zelime Elibol, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Undecided